CLINICAL TRIAL: NCT00001365
Title: NMDA Receptor Antagonist Treatment of Neurodegenerative Disease
Brief Title: Dextromethorphan for the Treatment of Parkinson's Disease and Similar Conditions of the Nervous System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930183; 93-N-0183
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2000-07

CONDITIONS: Neurodegenerative Disease; Parkinson's Disease
Keywords: Dextromethorphan; Dextrorphan; Glutamate Antagonist; Parkinson's Disease
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease | interventions — Dextromethorphan

INTERVENTIONS:
Drug: dextromethorphan

SUMMARY:
This study is designed to determine whether dextromethorphan, a drug commonly found in cough medicine, is beneficial and safe for the treatment of Parkinson's disease and other diseases that might share biochemical abnormalities with Parkinson's disease.

Patients with Parkinson's disease are missing the chemical neurotransmitter dopamine. This occurs as a result of destructive changes in an area of the brain responsible for making dopamine, the basal ganglia. Rhythmical muscular tremors, rigidity of movement, shuffling footsteps, droopy posture, and a mask-like expression on the face characterize Parkinson's disease.

Researchers believe that dextromethorphan may be able to safely modify psychomotor function of patients with Parkinson's Disease.

DETAILED DESCRIPTION:
The ability of the putative excitatory amino acid receptor antagonist, dextromethorphan, to modify psychomotor function safely in patients with neurodegenerative disease will be evaluated using a modified double-blind placebo-controlled design. Therapeutic activity will be rated at various doses by means of standard motor and cognitive performance scales. Safety will be assessed at frequent intervals by clinical observation and laboratory tests.

ELIGIBILITY:
Parkinson's disease or other neurodegenerative disorders in which excessive stimulation of central glutamatergic pathways is hypothesized.

Patients must be in good general health and have no history or clinical evidence of significant cardiac (including dysrhythmias), pulmonary, gastrointestinal, renal, hepatic, endocrine, hematological or psychiatric disease.

Patient must not evidence any disorder which in the opinion of the investigator imposes an unnecessary risk to the patient or compromises the scientific interpretation of the data.

Individuals of child bearing potential must practice appropriate methods of birth control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 1993-07; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Blanchet PJ, Papa SM, Metman LV, Mouradian MM, Chase TN. Modulation of levodopa-induced motor response complications by NMDA antagonists in Parkinson's disease. Neurosci Biobehav Rev. 1997 Jul;21(4):447-53. doi: 10.1016/s0149-7634(96)00038-3. PMID 9195602
- [Background] Verhagen Metman L, Blanchet PJ, van den Munckhof P, Del Dotto P, Natte R, Chase TN. A trial of dextromethorphan in parkinsonian patients with motor response complications. Mov Disord. 1998 May;13(3):414-7. doi: 10.1002/mds.870130307. PMID 9613730